CLINICAL TRIAL: NCT02439801
Title: Comparison of Effects of 3 Different PEEP Levels on Hemodynamic, Respiratory Mechanics and Elimination of Volatile Anesthetic Agent in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Comparison of Effects of PEEP Levels on Respiratory Mechanics in Patients Undergoing Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Umraniye Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gulsah Karaoren, MD, Umraniye Education and Research Hospital
Other Study IDs: GK5
Record Dates: First submitted 2015-05-03; First posted 2015-05-12 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Respiratory System Abnormalities
Keywords: PEEP; compliance; peak airway pressures
MeSH Terms: conditions — Respiratory System Abnormalities; Patient Compliance

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Compliance: Pulmonary compliance (or lung compliance) is a measure of the lung's ability to stretch and expand. In clinical practice it is separated into two different measurements, static compliance and dynamic compliance. Static lung compliance is the change in volume for any given applied pressure. Dynamic lung compliance is the compliance of the lung at any given time during actual movement of air.
  Effects of intra-operative PEEP 0, PEEP 5, PEEP 8 treatment on static and dynamic compliance levels will be investigate.
  Interventions: Procedure: PEEP 0; Procedure: PEEP 5; Procedure: PEEP 8
- Pulmonary Function tests: Pulmonary function testing has diagnostic and therapeutic roles and helps clinicians answer some general questions about patients with lung disease.
  Effects of intra-operative PEEP 0, PEEP 5, PEEP 8 treatment on pulmonary function test values will be investigate.
  Interventions: Procedure: PEEP 0; Procedure: PEEP 5; Procedure: PEEP 8
- volatil agent elimination time: Volatile anaesthetics are eliminated in the terminal phase via the lungs. A low blood:gas partition coefficient is therefore necessary for quick removal of the anaesthetic.
  Effects of intra-operative PEEP 0, PEEP 5, PEEP 8 treatment on volatil agent elimination time will be investigate.
  Interventions: Procedure: PEEP 0; Procedure: PEEP 5; Procedure: PEEP 8

INTERVENTIONS:
Procedure: PEEP 0 — 0 cmH2O positive end expiratory pressure
Procedure: PEEP 5 — 5 cmH2O positive end expiratory pressure
Procedure: PEEP 8 — 8 cmH2O positive end expiratory pressure

SUMMARY:
Laparoscopic cholecystectomy is accepted as gold standard in the management of cholelithiasis. Although laparoscopic procedures have many advantages,intra-abdominal CO2 insufflation can cause decreased lung volumes and compliance, increased airway resistance and impaired ventilation-perfusion ratio. In this study, investigators aim to investigate effects of intra-operative PEEP treatment at 3 distinct levels on respiratory dynamics and elimination time of volatile anesthetic agent.

DETAILED DESCRIPTION:
In the study, 75 ASA I-II patients aged 30-65 years will be randomized into 3 groups to receive 0 cmH2O PEEP (Group-1), 5 cmH2O PEEP (Group-2) and 8 cmH2O PEEP (Group-3) in PVC mode. In all patients underwent general anesthesia; hemodynamic parameters, Ppeak, Pplateau, compliance values as well as Fisevo/Fexpsevo ratio at 1 MAC and times from 1 MAC to 0.3 and 0.1 MAC will be recorded. In addition, preoperative and postoperative pulmonary function tests will be compared in all patients.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I-II
* BMI of 25-30
* patients scheduled to elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patients with ASA III, IV, V risk,
* Patients with comorbid diseases that may increase intra-abdominal pressure or pulmonary hypertension,
* Patients with renal and hepatic failure,
* Patients with pregnancy and
* Patients using bronchodilator or steroid were excluded.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who will undergo for elective laparoscopic cholecystectomy
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
levels of static-dynamic compliance with intra-operative PEEP treatment at 3 distinct levels | 1 month

SECONDARY OUTCOMES:
elimination time of volatile anesthetic agent with intra-operative PEEP treatment at 3 distinct levels | 1 month
levels of p peak and p plateau pressures with intra-operative PEEP treatment at 3 distinct levels | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Nurten Bakan, MD, Study Director — Unraniye training hospital
Locations (1):
- Istanbul Umraniye Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Karsten J, Heinze H, Meier T. Impact of PEEP during laparoscopic surgery on early postoperative ventilation distribution visualized by electrical impedance tomography. Minerva Anestesiol. 2014 Feb;80(2):158-66. Epub 2013 Jul 23. PMID 23877309
- [Result] Aydin V, Kabukcu HK, Sahin N, Mesci A, Arici AG, Kahveci G, Ozmete O. Comparison of pressure and volume-controlled ventilation in laparoscopic cholecystectomy operations. Clin Respir J. 2016 May;10(3):342-9. doi: 10.1111/crj.12223. Epub 2014 Nov 14. PMID 25307158
- [Result] Ozdilekcan C, Songur N, Berktas BM, Dinc M, Ucgul E, Ok U. Risk factors associated with postoperative pulmonary complications following oncological surgery. Tuberk Toraks. 2004;52(3):248-55. PMID 15351938